CLINICAL TRIAL: NCT06861023
Title: Review of the Literature and Retrospective, Single-centre Study of a Series of Patients Who Underwent Reconstruction After Complete Nail Resection.
Brief Title: Review of the Literature and Serie of Patients Who Underwent Reconstruction After Wide Local Excision of Nail Apparatus for Melanoma
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Chirplast01
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Plastic Surgery Procedures; Skin Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone extensive nail resection with reconstruction
  Interventions: Other: Patients who have undergone extensive nail resection with reconstruction

INTERVENTIONS:
Other: Patients who have undergone extensive nail resection with reconstruction — The investigators studied a population of 10 patients who underwent nail and nail matrix excision surgery as part of the treatment of subungual melanoma, as well as the reconstruction, the investigators opted for. The specific intervention of this study is based on late postoperative questions (after 3 months)
  Other Names: Excision of the nail apparatus with flap reconstruction or INTEGRA + skin graft.

SUMMARY:
Melanomas of the nail bed are often diagnosed at the locally advanced stage. The standard treatment was amputation of the finger or toe, but it has now been established that enlarged excision of the nail plate is sufficient under certain conditions. Reconstruction of the nail system can be performed by several techniques. Here, the investigators present a series of patients reconstructed by INTEGRA (dermal matrix) and skin graft

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone enlarged resection of the nail apparatus with immediate or delayed reconstruction in the setting of acral melanoma of the fingers or toes.

Exclusion Criteria:

* Patients who have amputation, opposition of the pateint to the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone melanoma surgery in the plastic surgery department of the Pasteur Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Functional and cosmetic patient satisfaction | 3 months minimum postoperative
  Scores AOFAS (feet)(score ranging from 0, maximum disability, to 90, no disability), Scores QUICK DASH(score ranging from 0, no disability, to 100, maximum disability) and Mayowrist score (hands)(score ranging from 0, maximum disability, to 100, no disability)

SECONDARY OUTCOMES:
Post-operative complications | 3 months minimum postoperative
  Presence or absence of Postoperative complications (inclusion cyst, nail spicule, need for repeat surgery).
Recurrence of the disease | 3 months minimum postoperative
  Recurrence of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France